CLINICAL TRIAL: NCT03675685
Title: A Phase 1, Open-Label Study to Assess the Safety and Pharmacokinetics of a Single Dose of CCH (3.36 mg) in Subjects With Edematous Fibrosclerotic Panniculopathy
Brief Title: Safety and Pharmacokinetics of a Single Dose of CCH (3.36 mg) in Subjects With EFP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-103
Record Dates: First submitted 2018-09-15; First posted 2018-09-18 (Actual); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Edematous Fibrosclerotic Panniculopathy
Keywords: Cellulite; Edematous Fibrosclerotic Panniculopathy; EFP
MeSH Terms: conditions — Cellulite | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CCH (Collagenase clostridium histolyticum) (Experimental)
  Interventions: Biological: CCH (collagenase clostridium histolyticum)

INTERVENTIONS:
Biological: CCH (collagenase clostridium histolyticum) — A single dose of 3.36 mg of CCH will be administered as subcutaneous injections (CCH 0.84 mg) per quadrant concurrently in 4 quadrants. A quadrant is defined as one of the following: left buttock, right buttock, left posterolateral thigh, or right posterolateral thigh.

SUMMARY:
This study will evaluate the safety and Pharmacokinetics (PK) of a single 3.36-mg dose of Collagenase Clostridium Histolyticum (CCH) in 4 quadrants concurrently, in subjects with Edematous fibrosclerotic panniculopathy (EFP).

This study will provide insight to the PK profile and safety of concurrent subcutaneous injections of CCH 0.84 mg/quadrant into 4 quadrants.

ELIGIBILITY:
Inclusion Criteria:

* No subject will be dosed until all eligibility criteria have been satisfied. In order to be eligible to participate in the study, subjects must meet the following criteria:

  1. Be a female ≥18 years of age.
  2. Have evidence of cellulite within 4 quadrants (a quadrant is defined as a left buttock, right buttock, left posterolateral thigh or right posterolateral thigh) as assessed by the Investigator using the Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) at the Screening visit; has a score of 2 (mild), 3 (moderate) or 4 (severe) as reported by the Investigator (CR-PCSS) in 4 quadrants at the Screening visit.
  3. Have a body mass index (BMI) between 20.0 and 35.0 kg/m^2, and intends to maintain stable body weight throughout the duration of the study (a variation of ≤10% from baseline body weight is permitted).
  4. Be willing to apply sunscreen to the dosing quadrants before each exposure to the sun while participating in the study (ie, screening through end of study).
  5. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile at screening.
  6. Have a negative pregnancy test at the Screening visit and on Day -1 at admission (before injection of study drug); and be using an effective contraception method (e.g., abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or double barrier control) for at least 1 menstrual cycle prior to study enrollment and for the duration of the study; or be menopausal defined as 12 months of amenorrhea in the absence of other biological or physiological causes, as determined by the Investigator; or post-menopausal for at least 1 year; or be surgically sterile (i.e., hysterectomy, bilateral oophorectomy, tubal ligation).
  7. Be willing and able to cooperate with the requirements of the study.
  8. Voluntarily sign and date an informed consent form approved by the Institutional Review Board/Independent Ethics Committee/Human Research Ethics Committee (IRB/IEC/HREC).

Exclusion Criteria:

* A subject will be excluded from study participation if she:

  1. Has any of the following systemic conditions:

     1. Coagulation disorder
     2. Evidence or history of malignancy (other than excised basal-cell carcinoma) unless there has been no recurrence in at least 5 years
     3. History of keloidal scarring or abnormal wound healing
     4. Concurrent diseases or conditions that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the subject's well-being. Any questions about concurrent diseases should be discussed with the Medical Monitor.
     5. Evidence of clinically significant abnormalities on physical examination, vital signs, electrocardiogram (ECG), or clinical laboratory values.
  2. Has any of the following local conditions in the areas to be treated:

     1. History of lower extremity thrombosis or post-thrombosis syndrome
     2. Vascular disorder (e.g., varicose veins) in areas to be treated
     3. Inflammation or active infection
     4. Active cutaneous alteration including rash, eczema, psoriasis, or skin cancer
     5. Has a tattoo located within 2 cm of the site of injection
  3. Requires the following concomitant medications before or during participation in the trial:

     a. Anticoagulant or antiplatelet medication or has received anticoagulant or antiplatelet medication (except for ≤150 mg aspirin daily) within 7 days before injection of study drug
  4. Has a positive test on a urine drug screen for drugs of abuse
  5. Has a history of drug or alcohol abuse
  6. Has used any of the following for the treatment of EFP on the legs or buttock within the timelines identified below or intends to use any of the following at any time during the course of the study:

     1. Liposuction within the treatment quadrants during the 12-month period before injection of study drug
     2. Injections (e.g., mesotherapy); radiofrequency device treatments; laser treatment; or surgery (including subcision and/or powered subcision) within the treatment quadrants during the 12-month period before injection of study drug
     3. Endermologie or similar treatments within the treatment quadrants during the 6-month period before injection of study drug
     4. Massage therapy within the treatment quadrants during the 3-month period before injection of study drug
     5. Creams (e.g., Celluvera™, TriLastin®) to prevent or mitigate EFP within the treatment quadrants during the 2-week period before injection of study drug
  7. Is presently nursing a baby or providing breast milk for a baby
  8. Intends to become pregnant during the study
  9. Intends to initiate an intensive sport or exercise program during the study
  10. Intends to initiate a weight reduction program during the study
  11. Has received an investigational drug or treatment within 30 days before injection of study drug
  12. Has a known systemic allergy to collagenase or any other excipient of study drug
  13. Has received any collagenase treatments at any time prior to treatment
  14. Has been a subject in a previous cellulite clinical trial of CCH: AUX-CC-830, AUX-CC-831, EN3835-102, EN3835-104, EN3835-201, EN3835-202, EN3835-205, EN3835-302, EN3835-303, EN3835-304, and/or EN3835-209.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saji Vijayan, MD, Study Director — Endo Pharmaceuticals
Locations (1):
- Endo Clinical Trial Site #1, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CCH (Collagenase Clostridium Histolyticum)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CCH (Collagenase Clostridium Histolyticum)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m^2)] | 29.94 (3.574)
Skin Category (Fitzpatrick Scale) [Count of Participants; unit: Participants]
  I (Pale White) | 0
  II (Fair) | 1
  III (Darker White) | 4
  IV (Light Brown) | 3
  V (Brown) | 1
  VI (Dark Brown or Black) | 3

OUTCOME MEASURES:

1. Primary Outcome: Plasma AUX-I and AUX-II Concentrations
Description: Determine if there is systemic exposure following a subcutaneous single dose of Collagenase clostridium histolyticum (CCH) (3.36 mg) as 12 injections per quadrant in 4 quadrants concurrently (0.84 mg per quadrant) in adult women with Edematous Fibrosclerotic Panniculopathy (EFP). There were no quantifiable levels of plasma AUX-I or AUX-II observed at any collection time point following subcutaneous injection of EN3835. As a result, no pharmacokinetic (PK) parameters were calculated.
Time Frame: Day 1 to Day 22
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | CCH (Collagenase Clostridium Histolyticum)
Number analyzed (Participants) | 12
mmol/L | NA (NA) — There were no quantifiable levels of plasma AUX-I or AUX-II observed at any collection time point following subcutaneous injection of EN3835- As a result, no Pharmacokinetic (PK) parameters were calculated.

2. Primary Outcome: Investigator CR-PCSS Rating
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) scores for each quadrant are based on the investigator's CR-PCSS evaluation done at the Screening visit (Baseline) and at End of Study (Day 22). CR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe). Negative change reflects an improvement in cellulite severity; positive change reflects a worsening in cellulite severity.
Time Frame: Day 1 to Day 22
Population: Cellulite Severity Population
Measure: Count of Participants; unit: Participants
Groups:
- Left Buttock; Right Buttock; Left Thigh; Right Thigh: CCH 0.84 mg/Area, 3.36 mg Total
Arm/Group | Left Buttock | Right Buttock | Left Thigh | Right Thigh
Number analyzed (Participants) | 11 | 11 | 11 | 11
Participants
  Screening (Baseline): None (0) | 0 | 0 | 0 | 0
  Screening (Baseline): Almost None (1) | 0 | 0 | 0 | 0
  Screening (Baseline): Mild (2) | 6 | 4 | 8 | 8
  Screening (Baseline): Moderate (3) | 4 | 6 | 3 | 3
  Screening (Baseline): Severe (4) | 1 | 1 | 0 | 0
  Day 22 (End of Study): None (0) | 0 | 0 | 0 | 0
  Day 22 (End of Study): Almost None (1) | 1 | 2 | 5 | 5
  Day 22 (End of Study): Mild (2) | 7 | 6 | 5 | 4
  Day 22 (End of Study): Moderate (3) | 3 | 1 | 1 | 2
  Day 22 (End of Study): Severe (4) | 0 | 2 | 0 | 0

3. Primary Outcome: Investigator CR-PCSS Change From Baseline
Description: Change from Baseline (Day 22 - Baseline). Baseline Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) scores for each quadrant are based on the investigator's CR-PCSS evaluation done at the Screening visit. CR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe). Negative change reflects an improvement in cellulite severity; positive change reflects a worsening in cellulite severity.
Time Frame: Day 1 to Day 22
Population: Cellulite Severity Population
Measure: Count of Participants; unit: Participants
Arm/Group | Left Buttock | Right Buttock | Left Thigh | Right Thigh
Number analyzed (Participants) | 11 | 11 | 11 | 11
Participants
  -4 | 0 | 0 | 0 | 0
  -3 | 0 | 0 | 0 | 0
  -2 | 0 | 1 | 1 | 0
  -1 | 5 | 4 | 5 | 7
  0 | 5 | 5 | 5 | 3
  +1 | 1 | 1 | 0 | 1
  +2 | 0 | 0 | 0 | 0

4. Primary Outcome: Investigator CR-PCSS Responder Analysis at End of Study
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) scores for each quadrant are based on the investigator's CR-PCSS evaluation at the end of study. CR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe). A 2-point responder is a participant with a reduction of cellulite severity by at least 2 severity levels from baseline to end of study (i.e., change from baseline CR-PCSS rating of -2, -3, or -4). A 1-point responder is a participant with a reduction of cellulite severity by at least 1 severity level from baseline to end of study (i.e., change from baseline CR-PCSS rating of -1, -2, -3, or -4).
Time Frame: Day 22
Population: Cellulite Severity Population
Measure: Count of Participants; unit: Participants
Arm/Group | Left Buttock | Right Buttock | Left Thigh | Right Thigh
Number analyzed (Participants) | 11 | 11 | 11 | 11
Participants
  2-point Responder: Yes | 0 | 1 | 1 | 0
  2-point Responder: No | 11 | 10 | 10 | 11
  1-point Responder: Yes | 5 | 5 | 6 | 7
  1-point Responder: No | 6 | 6 | 5 | 4

ADVERSE EVENTS:
Time Frame: All (serious and nonserious) AEs, from Day 1 up to Day 22
Description: All (serious and nonserious) AEs, whether elicited or observed during study visits or spontaneously reported by the participant, including events that occurred from the time the participant signed the study-specific consent form until completion of or discharge from the study.
Arm/Group | CCH (Collagenase Clostridium Histolyticum)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CCH (Collagenase Clostridium Histolyticum) (N=12)
Injection site bruising (General disorders) | 12
Injection site pain (General disorders) | 12
Injection site oedema (General disorders) | 4
Injection site swelling (General disorders) | 2
Chills (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site nodule (General disorders) | 1
Injection site pruritus (General disorders) | 1
Injection site warmth (General disorders) | 1
Pyrexia (General disorders) | 1
Headache (Nervous system disorders) | 2
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Drug withdrawal headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT03675685/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT03675685/SAP_001.pdf